CLINICAL TRIAL: NCT04930120
Title: TRANSCOV Cohort. An Epidemiological Study Assessing the Impact of Critically Ill COVID-19 Patients Long Distance Transfers Between Intensive Care Units
Brief Title: Assessing the Impact of COVID-19 Patients Long Distance Transfers Between Intensive Care Units
Acronym: TRANSCOV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ecole des Hautes Etudes en Santé Publique (Other)
Responsible Party: Principal Investigator, Olivier Grimaud, Head of the deparment Quantitative Methods in Public Health, Ecole des Hautes Etudes en Santé Publique
Other Study IDs: 20 CO 015 CZ
Record Dates: First submitted 2021-06-16; First posted 2021-06-18 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transferred group: The transferred group includes all severe COVID patients admitted in a French ICU ward and then transferred between the 03/13/2020 and 04/10/2020 to another ICU located outside the region of the initial ICU stay.
  Interventions: Other: Inter ICU long distance patient transfer
- Control group: The control group includes patients selected out of those whose entire ICU care has taken place in one of the hospitals which transferred patients. Up to 4 control patients will be selected for each transferred patient.

INTERVENTIONS:
Other: Inter ICU long distance patient transfer — Individual or grouped transportation between ICU of severely ill patients using ambulance, plane, helicopter, train or boat, with specialist medical assistance.
  Groups: Transferred group

SUMMARY:
The TRANSCOV cohort is a multicentre observational retrospective study aiming at assessing the health impact of extra regional transfers of critically ill COVID-19 patients.

DETAILED DESCRIPTION:
In spring 2020 four regions of France faced a surge of severe Coronavirus (COVID) patients which threatened to overflow local intensive care units (ICU) capacities. As an emergency response, between 03/13/2020 and 04/10/2020, an estimated 661 patients were transferred from overcrowded ICUs to other French regions and neighbouring countries. The study aims at assessing the impact of these inter-ICU transfers on the short and medium term physical and psychological outcomes in this population of severe COVID 19 patients.

All transferred patients between ICUs outside the origin region are invited to take part. For each transfer, up to four control patients will be selected among those admitted in the same ICU during the same period (+/-4 days of transfer date). Clinical data will be extracted from medical records and will include hemodynamic and respiratory parameters, as well as clinical severity scores before, during and after transfer. Data linkage with medico-administrative data will enrich the clinical database and allow follow-up up to one year after initial admission.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 patients diagnosed biologically or by imaging
* Admission in ICU between 03/13/2020 and 04/10/2020

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Severely ill COVID-19 patients
Sampling Method: Non-Probability Sample
Enrollment: 3060 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | 1 year
  Status alive or dead

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Grimaud, Ph.D., M.D., Principal Investigator — Ecole des Hautes Etudes en Santé Publique
Locations (1):
- EHESP, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided
undecided